CLINICAL TRIAL: NCT01584570
Title: The Effects of Dexmedetomidine and Tracheal Intubation on Heart Rate Variability and QTc Interval
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2011-0791
Record Dates: First submitted 2012-04-20; First posted 2012-04-25 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Anesthesia, General
Keywords: dexmedetomidine; heart rate variability; QTc interval
MeSH Terms: interventions — Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): fentanyl 1 mcg/kg before induction
  Interventions: Drug: 0.5 mcg/kg IV infusion for 10 min, 1.0 mcg/kg IV infusion for 10 min
- D 0.5 group (Experimental): Dexmedetomidine 0.5 ug/kg + Propofol + Sevoflurane+ Vecuronium
  Interventions: Drug: 0.5 mcg/kg IV infusion for 10 min, 1.0 mcg/kg IV infusion for 10 min
- D 1.0 group (Experimental): Dexmedetomidine 1.0 ug/kg + Propofol + Sevoflurane+ Vecuronium
  Interventions: Drug: 0.5 mcg/kg IV infusion for 10 min, 1.0 mcg/kg IV infusion for 10 min

INTERVENTIONS:
Drug: 0.5 mcg/kg IV infusion for 10 min, 1.0 mcg/kg IV infusion for 10 min — ECG monitoring for evaluation of QTc interval

SUMMARY:
The purpose of this study is to investigate effect of dexmedetomidine and tracheal intubation on heart rate variability and QTc interval.

ELIGIBILITY:
Inclusion Criteria:

* patient who are regarded as ASA class I
* age 20 to 60
* patient scheduled for Intubation for surgery

Exclusion Criteria:

* QTc interval > 440 ms
* arrythmia
* Patient who is taking a medicine which effects QTc interval
* HTN
* DM
* renal disease
* hepatic disease
* pregnant
* illiterate

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-01-01; Primary Completion 2013-12-23 (Actual); Study Completion 2013-12-23 (Actual)

PRIMARY OUTCOMES:
Change of QTc interval | T1 (at rest), T2 (5 min after dexmedetomidine infusion), T3 (just before intubation), T4(1 min after intubation), T5(2 min after intubation), T6(3min after intubation)
  T1- baseline, T2- to evaluate the effect of dexmedetomidine on QTc interval, T3- to evaluate QTc interval just before intubation, T4,5,6 - to evaluate QTc interval after intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea